CLINICAL TRIAL: NCT06105866
Title: Relationship of Preoperative Fasting With Tricuspid Annular Plane Systolic Excursion (TAPSE)
Brief Title: Relationship of Preoperative Fasting With Tricuspid Annular Plane Systolic Excursion
Acronym: (TAPSE)
Status: Enrolling by invitation | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, Assistant Professor, Aydin Adnan Menderes University
Other Study IDs: NCT093509350935
Record Dates: First submitted 2023-10-19; First posted 2023-10-30 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: The Relationship Between TAPSE Value and Volume
Keywords: Tricuspid Annular Plane Systolic Excursion; Preoperative Fasting; Right ventricular functions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients without Cardiac Disease: Patients between the ages of 18-75 with sinus rhythm, and without valvular disease, pulmonary hypertension, acute myocardial infarction, dilated, and hypertrophic cardiomyopathy will be included in the study.
  Interventions: Diagnostic Test: Tricuspid Annular Plane Systolic Excursion

INTERVENTIONS:
Diagnostic Test: Tricuspid Annular Plane Systolic Excursion — Transthoracic echocardiography will be performed on patients during hospitalization and preoperatively to investigate the relationship between preoperative fasting and right ventricular functions. This will be examined by looking at TAPSE

SUMMARY:
The aim of our study is to try to establish a relationship between preoperative fasting-related volume changes and tricuspid annular plane systolic excursion (TAPSE), and to determine whether there are changes in right ventricular functions due to preoperative fasting.

DETAILED DESCRIPTION:
TAPSE (Tricuspid Annular Plane Systolic Excursion) is a parameter that easily measures apex-base shortening and provides specific information about global right ventricular (RV) function. It is less dependent on optimal image quality and serves as an easily measurable criterion compared to other RV function measurements. In this study, one day before the operation, transthoracic echocardiography (TTE) will be conducted on fasting patients, and if the preoperative fasting duration is appropriate on the day of the surgery, TTE measurements will be repeated and recorded. The study aims to evaluate the relationship between TAPSE and volume and determine whether there are any changes in right ventricular functions due to preoperative fasting.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3
* The patient must be between 18 and 75 years old.
* Perioperative hydration has not been administered.
* Preoperative sedatives have not been given.
* There should be no known heart disease.

Exclusion Criteria:

* The patient being pregnant
* Post-cardiac surgery
* Severe pulmonary hypertension
* Severe valve disease
* Hypertrophic or dilated cardiomyopathy
* Presence of acute myocardial infarction
* Non-sinus rhythm

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery who have applied to Adnan Menderes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-11 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
The TAPSE value is related to volume | Patients who apply to our hospital for surgery within 6 months will be included in our study. Preoperative TAPSE measurements will be taken from the patients twice, first during admission and immediately before the operation
  We will measure FAC, S' velocity, TAPSE, and Myocardial Performance Index (MPI) derived from TDI to evaluate Right Ventricular (RV) systolic functions. To assess the RV diastolic function, we will measure Tricuspid E and A wave velocities, E/A ratio, and E' velocity. TAPSE will be calculated by placing an M-mode cursor along the Tricuspid Annulus and measuring the longitudinal excursion during peak systole

CONTACTS AND LOCATIONS:
Locations (1):
- Sevil Gulasti, Aydin, Zafer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the results of the statistical analysis of all collected data will be shared.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Lee S, Kamdar F, Madlon-Kay R, Boyle A, Colvin-Adams M, Pritzker M, John R. Effects of the HeartMate II continuous-flow left ventricular assist device on right ventricular function. J Heart Lung Transplant. 2010 Feb;29(2):209-15. doi: 10.1016/j.healun.2009.11.599. PMID 20113911
- [Background] Gullupinar B, Saglam C, Koran S, Turhan A, Unluer EE. The role of mitral annular plane systolic excursion in prediction of acute blood loss in healthy voluntary blood donors. J Ultrason. 2022 Feb 8;22(88):e33-e38. doi: 10.15557/JoU.2022.0006. eCollection 2022 Mar. PMID 35449700
- [Background] Zhang H, Wang X, Chen X, Zhang Q, Liu D. Tricuspid annular plane systolic excursion and central venous pressure in mechanically ventilated critically ill patients. Cardiovasc Ultrasound. 2018 Aug 7;16(1):11. doi: 10.1186/s12947-018-0130-2. PMID 30081914
- [Background] Newman K, Wilson R, Roberts JM, Mayo JR, Mohamed Ali AA, Brunner N, Sedlic A. Tricuspid annular plane systolic excursion for the evaluation of right ventricular function in functional cardiac CT compared to MRI. Clin Radiol. 2021 Aug;76(8):628.e1-628.e7. doi: 10.1016/j.crad.2021.02.018. Epub 2021 Apr 18. PMID 33879320